CLINICAL TRIAL: NCT07144748
Title: 68Ga-NYM096 PET/CT: Tracer Uptake in Various Kinds of Cancer
Brief Title: 68Ga-NYM096 PET/CT in Various Kinds of Cancer
Acronym: NYCRVT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: K8490
Record Dates: First submitted 2025-08-11; First posted 2025-08-27 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-07

CONDITIONS: Cancer
Keywords: 68Ga-NYM096; PET/CT; cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-NYM096 PET/CT (Experimental): Each patient will receive one dose of 68Ga-NYM096 by intravenous route. Dedicated whole-body PET/CT imaging will be performed.
  Interventions: Other: 68Ga-NYM096 PET/CT

INTERVENTIONS:
Other: 68Ga-NYM096 PET/CT — Participants will be administered a single, intravenous bolus of 68Ga-NYM096 The recommended administered activity of 68Ga-NYM096 is 1.8-2.2 MBq per kilogram bodyweight, subject to variation that may be required owing to variable elution efficiencies obtained during the lifetime of the 68Ga / 68Ga generator. The CT and PET imaging session will begin approximately 45 to 75 minutes after 68Ga-NYM096 administration.

SUMMARY:
This is a prospective, single-center study aimed at evaluating the uptake characteristics of 68Ga-NYM096 PET/CT in various kinds of tumors including primary and metastatic lesions. Based on image analysis, this study will assess the uptake of various kinds of tumors using 68Ga-NYM096 PET/CT. The findings will provide critical insights into the tumor uptake on 68Ga-NYM096 PET/CT to identify the most promising indications for future application.

DETAILED DESCRIPTION:
This is a prospective, single-center study designed to evaluate the uptake characteristics of 68Ga-NYM096 PET/CT in various kinds of tumors including primary and metastatic lesions. Each patient will receive a single intravenous dose of 68Ga-NYM096, followed by dedicated whole-body PET/CT imaging. 68Ga-NYM096 PET/CT scans were requested by referring physicians according to individual clinical indications that were considered insufficiently covered by 18F-FDG PET/CT or other imaging modalities.

Quantitative analyses will be applied to assess the uptake of 68Ga-NYM096 in primary and metastatic lesions in different tumor types, including lesion number, SUVmax (40% isocontour), tumor-to-background ratio (TBR).

120 patients with histopathologically proven primary tumors or metastases or radiologically unequivocal metastatic lesions of histologically proven primary tumors will be recruited in Peking Union Medical College Hospital. This study will be conducted according to local regulations and laws, the ethical principles that have their origin in the Declaration of Helsinki, and the principles of Good Clinical Practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 y
2. Histopathologically confirmed cancer (histopathologically proven primary tumors or metastases or radiologically unequivocal metastatic lesions of histologically proven primary tumors)
3. Expected survival of at least 3 months
4. ECOG ≤ 2
5. Written informed consent provided for participation in the trial
6. In the opinion of investigator, willing and able to comply with required study procedures.

Exclusion Criteria:

1. On VEGF TKI treatment less than 1 week before 68Ga-NYM096 PET/CT. TKI is known to affect girentuximab binding in patients with ccRCC and is expected to have the same effect on 68Ga-NYM096. If patients were on VEGF TKI treatment, such as sunitinib, sorafenib, cabozantinib, pazopanib, or lenvatinib, a washout of one week before 68Ga-NYM096 PET/CT is required.
2. Intercurrent medical condition that renders the patient ineligible for the procedures.
3. Pregnancy or breastfeeding.
4. Severe claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Uptake characteristics (quantitative analysis) of tumor lesions including primary and metastatic lesions identified on 68Ga-NYM096 PET/CT | From study completion to 1 month after completion
  For tumor lesions, the tracer uptake is quantified using maximal and mean standard uptake value by drawing a 3-dimensional region of interest (ROI) over the lesion using a threshold of 40% SUVmax. Tumor-to-background ratios (TBRs) should also be evaluated. Adjacent normal tissue is the preferred background tissue. If not available, the blood pool should be designated as background tissue.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing 100730, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Available upon request
Supporting Information: Study Protocol
Time Frame: Within 2 years after the publication of the main results